CLINICAL TRIAL: NCT05208970
Title: Genetic Diversity of Cryptosporidium Species Infecting Human in Sohag Governorate
Brief Title: Cryptosporidium Species in Sohag Governorate
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salwa Gamal Ahmed Omran, assistant lecturer of medical parasitology, Sohag University
Other Study IDs: Soh-Med-22-01-12
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cryptosporidiosis
MeSH Terms: conditions — Cryptosporidiosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cryptosporidium species are increasingly recognized as important enteric pathogens that infect a broad range of hosts including human, domestic and wild animals worldwide, causing asymptomatic or mild-to-severe gastrointestinal disease in their host species.

There are 38 species of Cryptosporidium that have been described, going from amphibian parasites to mammals ones, with over 40 genotypes infecting mammals, although Cryptosporidium parvum and Cryptosporidium hominis are the two species predominantly reported in human infections. In Cairo and Sharkyia governorates in Egypt, Cryptosporidium is a common intestinal parasite among children, especially in diarrheic, preschool-aged children, with a predominance of C. hominis indicates anthroponotic rather than zoonotic transmission. Also in the sohag governorate, Cryptosporidium infection is a common intestinal parasite, as in the last five years its prevalence about 35% but there is no study clarify predominant genotype of Cryptosporidium in sohag.

ELIGIBILITY:
Inclusion Criteria:

1. Age: any age
2. Sex: male -female
3. Residence: rural-urban
4. Animal contact.
5. Immune status: immunocompetent - immunocompromised
6. Clinical manifestations: diarrhea -abdominal pain- fever- vomiting.

Exclusion Criteria:

* patients taking treatment for cryptosporidiosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients at Sohag University Hospital will be sampled.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
estimate the prevalence and clarify the species and genotypes/subtypes of Cryptosporidium spp. in sohag. | 24 weeks

SECONDARY OUTCOMES:
clarify the relationship of them in a phylogenetic context and to provide additional information on the molecular epidemiology of this parasite in our locality | 24 weeks
clarify the predominant clinical manifestation of each genotypes/subtypes of Cryptosporidium spp | 24 weeks
clarify the relationship between genotypes/subtypes of Cryptosporidium spp. and different risk factors. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benamrouz S, Guyot K, Gazzola S, Mouray A, Chassat T, Delaire B, Chabe M, Gosset P, Viscogliosi E, Dei-Cas E, Creusy C, Conseil V, Certad G. Cryptosporidium parvum infection in SCID mice infected with only one oocyst: qPCR assessment of parasite replication in tissues and development of digestive cancer. PLoS One. 2012;7(12):e51232. doi: 10.1371/journal.pone.0051232. Epub 2012 Dec 13. PMID 23272093
- [Background] Ryan U, Zahedi A, Paparini A. Cryptosporidium in humans and animals-a one health approach to prophylaxis. Parasite Immunol. 2016 Sep;38(9):535-47. doi: 10.1111/pim.12350. PMID 27454991
- [Background] Kvac M, Havrdova N, Hlaskova L, Dankova T, Kandera J, Jezkova J, Vitovec J, Sak B, Ortega Y, Xiao L, Modry D, Chelladurai JR, Prantlova V, McEvoy J. Cryptosporidium proliferans n. sp. (Apicomplexa: Cryptosporidiidae): Molecular and Biological Evidence of Cryptic Species within Gastric Cryptosporidium of Mammals. PLoS One. 2016 Jan 15;11(1):e0147090. doi: 10.1371/journal.pone.0147090. eCollection 2016. PMID 26771460
- [Background] Mohammad SM, Ali MS, Abdel-Rahman SA, Moustafa RA, Sarhan MH. Genotyping of Cryptosporidium species in children suffering from diarrhea in Sharkyia Governorate, Egypt. J Infect Dev Ctries. 2021 Oct 31;15(10):1539-1546. doi: 10.3855/jidc.14367. PMID 34780378